CLINICAL TRIAL: NCT04988308
Title: A Phase 2a/2b, Multicenter, Randomized, Placebo and Active Comparator-controlled, Double-Blind, Dose-ranging Study to Evaluate the Safety and Efficacy of Bermekimab (JNJ-77474462) for the Treatment of Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study of Bermekimab for the Treatment of Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: LYRA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been prematurely terminated as the Interim Analysis 1 efficacy results met the prespecified futility criteria related to the primary endpoint.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109063; 2020-002607-19 (EudraCT Number); 77474462HDS2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-30; First posted 2021-08-03 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bermekimab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 (Group 1): Placebo (Placebo Comparator): Participants will receive placebo subcutaneously (SC) at Week 0 through Week 15. At Week 16, participants will cross over to receive bermekimab dose 1 SC every week thereafter through Week 31.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part 1 (Group 2): Adalimumab (Active Comparator): Participants will receive adalimumab 160 milligrams (mg) SC at Week 0, placebo SC at Week 1, followed by adalimumab 80 mg SC and placebo SC at Weeks 2 and 3. Participants will then receive adalimumab 40 mg SC and placebo SC at Week 4 and every week thereafter through Week 31.
  Interventions: Drug: Adalimumab; Drug: Placebo
- Part 1 (Group 3): Bermekimab Dose 1 (Experimental): Participants will receive bermekimab dose 1 SC and placebo SC at Week 0, followed by bermekimab dose 1 SC at Week 1 and every week thereafter through Week 31.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part 2 (Group 1): Placebo (Placebo Comparator): Participants will receive placebo SC from Week 0 through Week 11. At Week 12, participants will cross over to receive bermekimab dose 1 SC weekly through Week 31.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part 2 (Group 2): Bermekimab Dose 1 (Experimental): Participants will receive bermekimab dose 1 SC at Week 0 and every week thereafter through Week 31.
  Interventions: Drug: Bermekimab
- Part 2 (Group 3): Bermekimab Dose 1 (Experimental): Participants will receive bermekimab dose 1 SC at Week 0 and every week thereafter through Week 11. From Week 12, participants will receive bermekimab dose 1 SC every other week thereafter through Week 30. During weeks in which bermekimab is not administered, participants will receive placebo SC through Week 31.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part 2 (Group 4): Bermekimab Dose 2 (Experimental): Participants will receive bermekimab dose 2 SC and placebo SC at Week 0 and every week thereafter through Week 11. From Week 12, participants will receive bermekimab dose 2 SC and placebo SC every other week thereafter through Week 30. During weeks in which bermekimab is not administered, participants will receive placebo SC through Week 31.
  Interventions: Drug: Bermekimab; Drug: Placebo

INTERVENTIONS:
Drug: Bermekimab — Bermekimab will be administered subcutaneously.
  Other Names: JNJ-77474462
  Arms: Part 1 (Group 1): Placebo; Part 1 (Group 3): Bermekimab Dose 1; Part 2 (Group 1): Placebo; Part 2 (Group 2): Bermekimab Dose 1; Part 2 (Group 3): Bermekimab Dose 1; Part 2 (Group 4): Bermekimab Dose 2
Drug: Adalimumab — Adalimumab will be administered subcutaneously.
  Arms: Part 1 (Group 2): Adalimumab
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Part 1 (Group 1): Placebo; Part 1 (Group 2): Adalimumab; Part 1 (Group 3): Bermekimab Dose 1; Part 2 (Group 1): Placebo; Part 2 (Group 3): Bermekimab Dose 1; Part 2 (Group 4): Bermekimab Dose 2

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of bermekimab in participants with moderate to severe Hidradenitis Suppurativa (HS).

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic skin disease of unclear etiology that affects 1 percent (%) to 4% of the general population. JNJ-77474462 (bermekimab) is a recombinant human immunoglobulin G1 kappa (IgG1k) monoclonal antibody (mAb) that binds with high affinity and selectivity for human interleukin-1 alpha (IL-1 alpha) and is an effective blocker of IL-1 alpha biological activity. IL-1 alpha is a key mediator of sterile inflammatory responses. Skin is a significant reservoir of preformed IL-1 alpha, and it has been postulated that IL-1 alpha may play a role in the pathophysiology of multiple inflammatory skin disorders, including HS. Part 1 of this study contains 4 study periods: up to 6 weeks screening period (Period 1), 16-week placebo-controlled period (Period 2), 16-week cross over period (Period 3), and 4-week safety follow-up (Period 4). Part 2 of this study also contains 4 study periods: up to 6 weeks screening period (Period 1), 12-week placebo-controlled period (Period 2), 20-week cross over period (Period 3), and 4-week safety follow up (Period 4). Safety will be assessed by adverse events (AEs), serious adverse event (SAEs), physical examinations, vital signs, electrocardiograms, clinical safety laboratory assessments, allergic reaction, injection-site reactions, and tuberculosis evaluations. The total duration of study participation will be up to 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have hidradenitis suppurativa (HS) for at least 1 year (365 days) prior to the baseline visit as determined by the investigator through participant interview and/or review of the medical history
* Have Hurley Stage II or Hurley Stage III HS as determined by the investigator at screening and baseline visits
* Have HS lesions present in at least 2 distinct anatomic areas (examples include but are not limited to left and right axilla; or left axilla and left inguinocrural fold) at screening and baseline visits
* Have a total abscess and inflammatory nodule (AN) count of greater than or equal to (>=) 5 at the screening and baseline visit
* Agree not to receive a live virus or live bacterial vaccination during the study and for 90 days after the last administration of study intervention

Exclusion Criteria:

* Has a current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (that is, unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months
* Has or has had herpes zoster within the 2 months before screening
* Has a transplanted organ (with exception of a corneal transplant greater than [>] 3 months before the first administration of study intervention)
* Has known allergies, hypersensitivity, or intolerance to bermekimab or adalimumab or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (54):
- United States (22):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - Renstar Medical Research, Ocala, Florida
  - Forcare Clinical Research, Inc., Tampa, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Allcutis Research, Beverly, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Clarkston Dermatology & Vein Center, PLLC, Clarkston, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - JDR Dermatology Research, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - Wright State Physicians Health Center, Dayton, Ohio
  - Penn State Milton S. Hershey Medical Ctr., Hershey, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Arlington Center for Dermatology, Arlington, Texas
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Australia (4):
  - Clinical Trials SA Pty Ltd, Campbelltown
  - Holdsworth House, Darlinghurst
  - Sinclair Dermatology, East Melbourne
  - Veracity Clinical Research, Woolloongabba
- Canada (4):
  - SimcoMed Health Ltd, Barrie, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Centre De Recherche Dermatologique Du Quebec Metropolitan, Québec, Quebec
- Germany (6):
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Universitaetsklinik Erlangen, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitaets-Hautklinik Kiel, Kiel
  - Universitaetsmedizin Mainz, Mainz
  - Universitätsklinikum Würzburg, Würzburg
- Japan (5):
  - Fukuoka University Hospital, Fukuoka
  - Nagoya City University Hospital, Nagoya
  - University of the Ryukyus Hospital, Nakagami-gun
  - Meiwa Hospital, Nishinomiya
  - Takagi Dermatology Clinic, Obihiro-shi
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (4):
  - Centrum Medyczne Dermoklinika, Lódź
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Centrum Medyczne Matusiak w CITYCLINICPrzychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw
  - Wromedica, Wroclaw
- Spain (7):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Provincial de Pontevedra, Pontevedra
  - Hosp. de Manises, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per change in planned analysis, Part 2 of this study was not conducted due to early termination because interim analysis 1 efficacy results met the prespecified futility criteria related to the primary endpoint. Hence, data for Part 2 and some secondary efficacy outcome measures (Parts 1 and 2) were not reported in this results summary.
Groups:
- Part 1: Placebo (Week 0-16): Participants received placebo as subcutaneous (SC) injection from Week 0 through Week 15 and then participants received bermekimab 1050 milligrams (mg) as SC injection at Week 16 in Part 1.
- Part 1: Bermekimab (Week 0-36): Participants received bermekimab 1050 mg (3*350 mg) and 1 placebo as SC injection at Week 0 followed by bermekimab 1050 mg (3*350 mg) as SC injection at Week 1 and every week thereafter through Week 16 in Part 1. Participants who received bermekimab 1050 mg (3*350 mg) at Week 16 entered into active treatment + safety follow up (FU) period and received bermekimab 1050 mg as SC injection weekly through Week 36 in Part 1.
- Part 1: Adalimumab (Week 0-16): Participants received adalimumab 160 mg (4*40 mg) as SC injection at Week 0 and 3 placebo SC injections at Week 1 followed by adalimumab 80 mg (2*40 mg) as SC injection at Week 2 and 3 placebo SC injections at Week 3. Participants received adalimumab 40 mg (1*40 mg) SC injection and 2 placebo SC injections at Week 4 and every week thereafter through Week 16 in Part 1.
- Part 1: Placebo Then Bermekimab (Week 17-36): Participants who received placebo during placebo controlled period and then received bermekimab 1050 mg (3*350 mg) at Week 16 entered into active treatment + safety follow up (FU) period and received bermekimab 1050 mg as SC injection weekly through Week 31 in Part 1. All participants were followed for safety through Week 36.
- Part 1: Bermekimab (Week 17-36): Participants who received bermekimab 1050 mg at Week 16 during placebo controlled period entered into active treatment + safety FU period and continued to receive bermekimab 1050 mg (3*350 mg) as SC injection every week thereafter through Week 31. All participants were followed for safety through Week 36.
- Part 1: Adalimumab (Week 17-36): Participants who received adalimumab 40 mg as SC injection during placebo controlled period entered into active treatment period and continued to receive adalimumab 40 mg as SC injection and 2 placebo SC injections weekly through Week 31 in Part 1. All participants were followed for safety through Week 36.
Period: Placebo Controlled Period (Weeks 0-16)
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-36) | Part 1: Adalimumab (Week 0-16) | Part 1: Placebo Then Bermekimab (Week 17-36) | Part 1: Bermekimab (Week 17-36) | Part 1: Adalimumab (Week 17-36)
Started | 50 | 51 | 50 | 0 | 0 | 0
Full- Analysis Set (FAS) | 35 | 35 | 35 | 0 | 0 | 0
Completed | 28 | 30 | 28 | 0 | 0 | 0
Not Completed | 22 | 21 | 22 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Other | 10 | 9 | 14 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 6 | 4 | 3 | 0 | 0 | 0
Period: Active Treatment+Safety F-U (Week 17-36)
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-36) | Part 1: Adalimumab (Week 0-16) | Part 1: Placebo Then Bermekimab (Week 17-36) | Part 1: Bermekimab (Week 17-36) | Part 1: Adalimumab (Week 17-36)
Started | 0 | 0 | 0 | 28 (All participants who completed placebo-controlled period entered in active treatment + safety follow-up period.) | 30 (All participants who completed placebo-controlled period entered in active treatment + safety follow-up period.) | 28 (All participants who completed placebo-controlled period entered in active treatment + safety follow-up period.)
Completed | 0 | 0 | 0 | 7 | 9 | 10
Not Completed | 0 | 0 | 0 | 21 | 21 | 18
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 3 | 1
Not completed — Other | 0 | 0 | 0 | 10 | 10 | 14
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 5 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-36) | Part 1: Adalimumab (Week 0-16) | Total
Number analyzed (Participants) | 50 | 51 | 50 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12.55) | 36.7 (9.67) | 35.7 (12.2) | 36.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 28 | 83
  Male | 25 | 21 | 22 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 4 | 17
  Not Hispanic or Latino | 38 | 42 | 41 | 121
  Unknown or Not Reported | 5 | 3 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 10 | 3 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 8 | 17
  White | 32 | 37 | 32 | 101
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 5 | 2 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 1 | 4 | 4 | 9
  CANADA | 4 | 5 | 5 | 14
  GERMANY | 12 | 10 | 10 | 32
  JAPAN | 5 | 2 | 1 | 8
  NETHERLANDS | 0 | 1 | 0 | 1
  POLAND | 5 | 7 | 8 | 20
  SPAIN | 2 | 2 | 1 | 5
  UNITED STATES | 21 | 20 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Who Achieved Hidradenitis Suppurativa Clinical Response-50 (HiSCR50) at Week 16
Description: HiSCR50 was defined as at least 50 percent (%) reduction in total abscess and inflammatory nodule counts (AN count) with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 16
Population: The full analysis set (FAS) included all randomized participants who received at least one administration of study intervention.
Measure: Number; unit: Percentage of participants
Groups:
- Part 1: Bermekimab (Week 0-16): Participants received bermekimab 1050 mg (3*350 mg) and 1 placebo as SC injection at Week 0 followed by bermekimab 1050 mg (3*350 mg) as SC injection at Week 1 and every week thereafter through Week 16 in Part 1.
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 35 | 35 | 35
Percentage of participants | 37.1 | 37.1 | 57.1

2. Secondary Outcome: Part 1: Percentage of Participants Who Achieved HiSCR75 at Week 16
Description: HiSCR75 was defined as at least 75% reduction in total abscess and inflammatory nodule counts (AN count) with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 16
Population: The FAS included all randomized participants who received at least one administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 35 | 35 | 35
Percentage of participants | 25.7 | 25.7 | 40.0

3. Secondary Outcome: Part 1: Percentage of Participants Who Achieved HiSCR90 at Week 16
Description: HiSCR90 was defined as at least 90% reduction in total abscess and inflammatory nodule counts (AN count) with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 16
Population: The FAS included all randomized participants who received at least one administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 35 | 35 | 35
Percentage of participants | 14.3 | 17.1 | 22.9

4. Secondary Outcome: Part 1: Change From Baseline in the Abscess and Inflammatory Nodule (AN) Count at Week 16
Description: Change from baseline in the AN count as Week 16 was reported. Abscess and inflammatory nodule were counted for the hidradenitis suppurativa (HS) affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Baseline, Week 16
Population: The FAS included all randomized participants who received at least one administration of study intervention. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Abscess and inflammatory nodule
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 28 | 29 | 28
Abscess and inflammatory nodule | -4.50 (5.088) | -5.31 (8.594) | -7.25 (4.774)

5. Secondary Outcome: Part 1: Change From Baseline in Number of Abscess at Week 16
Description: Change from baseline in number of abscess at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Abscess
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 28 | 29 | 28
Abscess | -0.86 (1.900) | -0.83 (3.071) | -1.46 (2.333)

6. Secondary Outcome: Part 1: Change From Baseline in Number of Draining Fistula at Week 16
Description: Change from baseline in number of draining fistula at Week 16 was reported. Draining fistula was defined as fistulas that drain serous or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: fistulas
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 28 | 29 | 28
fistulas | -0.04 (1.915) | -1.00 (1.626) | -0.96 (1.575)

7. Secondary Outcome: Part 1: Change From Baseline in Number of Inflammatory Nodules at Week 16
Description: Change from baseline in number of inflammatory nodules at Week 16 was reported. Inflammatory nodules arise from inflamed blood vessels (vasculitis) or adipose tissue (panniculitis).
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: inflammatory nodules
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 28 | 29 | 28
inflammatory nodules | -3.64 (5.258) | -4.48 (7.689) | -5.79 (4.306)

8. Secondary Outcome: Part 1: Change From Baseline in International Hidradenitis Suppurativa Severity Score (IHS4) at Week 16
Description: IHS4 was a dynamic severity assessment of HS. IHS4 score was arrived at by the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease. Higher scores indicate more severity.
Time Frame: Baseline up to Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 28 | 29 | 28
scores on a scale | -5.5 (10.38) | -10.14 (13.36) | -12.6 (9.15)

9. Secondary Outcome: Part 1: Percentage of Participants With Hidradenitis Suppurativa-Investigator's Global Assessment (HS-IGA) Score of Inactive (0), Almost Inactive (1), or Mild Activity (2) and With at Least 2-grade Improvement Relative to Baseline at Week 16
Description: The HS-IGA documents the investigator's assessment of the participant's HS at a given timepoint. The anatomic region with the most severe HS activity at the baseline was evaluated for erythema, drainage, and pain and/or tenderness to palpation for each participant. The participant's HS was assessed as inactive (0), almost inactive (1), mild activity (2), moderate activity (3), or severe activity (4). A higher score indicates more severe disease. Percentage of participants with HS-IGA score of inactive (0), almost inactive (1), or mild activity (2) and with at least 2-grade improvement relative to baseline at Week 16 were reported.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 35 | 35 | 34
Percentage of participants
  HS-IGA scores of inactive (0) | 11.4 | 17.1 | 20.6
  HS-IGA scores of inactive (0) or almost active (1) | 25.7 | 25.7 | 38.2
  HS-IGA scores of inactive (0), or or almost active (1), or mild activity (2) | 28.6 | 28.6 | 38.2

10. Secondary Outcome: Part 1: Change From Baseline in Hidradenitis Suppurativa (HS)-Related Pain Symptom Score in the Past 24 Hours Based on Hidradenitis Suppurativa Symptom Diary (HSSD) Questionnaire at Week 16
Description: HSSD is a 7-item patient self-reported questionnaire that assesses 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms have a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours with a score range from 0 (no symptom experience) to 10 (worst possible symptom experience). A total symptom score also ranged from 0 (no symptom) to 10 (worst possible symptom), was derived by averaging the 5 individual scale scores that utilize the past 7-day recall period. Change from baseline in HS-related pain symptom score in the past 24 hours based on HSSD was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-16) | Part 1: Adalimumab (Week 0-16)
Number analyzed (Participants) | 20 | 22 | 20
scores on a scale | -1.00 (2.461) | -0.41 (2.374) | -1.96 (2.326)

11. Secondary Outcome: Serum Concentration of Bermekimab
Description: Serum concentration of bermekimab was reported. As per planned analysis, this outcome measure was analyzed in a single arm for participants who received bermekimab from Week 0 to Week 36.
Time Frame: Weeks 0, 1, 4, 8, 12, 16, 20, 24, 28, 32, 36
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of bermekimab and had at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at each specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Part 1: Bermekimab (Week 0-36)
Number analyzed (Participants) | 50
micrograms per milliliter (mcg/mL)
  Week 0 | 0.00 (0.000)
  Week1: number analyzed (Participants) | 47
  Week1 | 51.36 (20.354)
  Week 4: number analyzed (Participants) | 36
  Week 4 | 78.46 (43.897)
  Week 8: number analyzed (Participants) | 22
  Week 8 | 73.14 (37.583)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 72.45 (39.185)
  Week 16: number analyzed (Participants) | 14
  Week 16 | 61.81 (42.092)
  Week 20: number analyzed (Participants) | 12
  Week 20 | 74.68 (59.300)
  Week 24: number analyzed (Participants) | 10
  Week 24 | 89.75 (50.940)
  Week 28: number analyzed (Participants) | 7
  Week 28 | 66.30 (57.219)
  Week 32: number analyzed (Participants) | 4
  Week 32 | 34.53 (36.160)
  Week 36: number analyzed (Participants) | 4
  Week 36 | 4.63 (7.576)

12. Secondary Outcome: Number of Participants With Antibodies to Bermekimab
Description: Number of participants with antibodies to bermekimab was reported. As per planned analysis, this outcome measure was analyzed in a single arm for participants who received bermekimab from Week 0 to Week 36.
Time Frame: From baseline up to Week 36
Population: The immunogenicity analysis set included all participants who received at least 1 dose of bermekimab and who had at least 1 sample obtained after their first dose of bermekimab for the detection of antibodies to bermekimab.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Bermekimab (Week 0-36): Participants received bermekimab 1050 mg (3*350 mg) and 1 placebo as SC injection at Week 0 followed by bermekimab 1050 mg (3*350 mg) as SC injection at Week 1 and every week thereafter through Week 16 in Part 1. Participants who received bermekimab 1050 mg (3*350 mg) at Week 16 entered into active treatment + safety follow up (FU) period and received bermekimab 1050 mg as SC injection weekly through Week 31 in Part 1. All participants were followed for safety through Week 36.
Arm/Group | Part 1: Bermekimab (Week 0-36)
Number analyzed (Participants) | 51
Participants | 16

ADVERSE EVENTS:
Time Frame: Part 1: Placebo Controlled Period: From Week 0 to Week 16; Active Treatment + Safety Follow-up Period: From Week 17 to Week 36
Description: The safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Part 1: Placebo (Week 0-16) | Part 1: Bermekimab (Week 0-36) | Part 1: Adalimumab (Week 0-16) | Part 1: Placebo Then Bermekimab (Week 17-36) | Part 1: Bermekimab (Week 17-36) | Part 1: Adalimumab (Week 17-36)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 1/50 | 0/28 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/51 | 4/50 | 0/28 | 1/30 | 1/28
Other Adverse Events (participants affected / at risk) | 21/50 | 31/51 | 22/50 | 12/28 | 12/30 | 11/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (Week 0-16) (N=50) | Part 1: Bermekimab (Week 0-36) (N=51) | Part 1: Adalimumab (Week 0-16) (N=50) | Part 1: Placebo Then Bermekimab (Week 17-36) (N=28) | Part 1: Bermekimab (Week 17-36) (N=30) | Part 1: Adalimumab (Week 17-36) (N=28)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Skin Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (Week 0-16) (N=50) | Part 1: Bermekimab (Week 0-36) (N=51) | Part 1: Adalimumab (Week 0-16) (N=50) | Part 1: Placebo Then Bermekimab (Week 17-36) (N=28) | Part 1: Bermekimab (Week 17-36) (N=30) | Part 1: Adalimumab (Week 17-36) (N=28)
Nausea (Gastrointestinal disorders) | 1 | 5 | 4 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3 | 2 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 3 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 16 | 3 | 5 | 1 | 0
Injection Site Pruritus (General disorders) | 0 | 9 | 1 | 5 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Covid-19 (Infections and infestations) | 5 | 4 | 3 | 1 | 2 | 4
Nasopharyngitis (Infections and infestations) | 2 | 4 | 4 | 2 | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4 | 3 | 1 | 3 | 2
C-Reactive Protein Increased (Investigations) | 1 | 3 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 6 | 6 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 6 | 3 | 1 | 0 | 4 | 1

LIMITATIONS AND CAVEATS:
As per change in planned analysis, Part 2 and some secondary efficacy analysis of Part 1 in this study was not conducted due to early termination because interim analysis 1 efficacy results met the prespecified futility criteria related to the primary endpoint. Hence, data for Part 2 and some secondary efficacy outcome measures (Parts 1 and 2) were not collected in this results summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04988308/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT04988308/SAP_001.pdf